CLINICAL TRIAL: NCT05414604
Title: Calculating the Volume of the Paravertebral Space With 3D Computerized Tomography
Brief Title: Calculating the Volume of the Paravertebral Space
Status: Completed | Type: Observational
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Can AKSU, MD, Principal investigator., Kocaeli University
Other Study IDs: GOKAEK-2021/16.20
Record Dates: First submitted 2022-06-04; First posted 2022-06-10 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Vertebral Disc Degenerative Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PV group: Patients who had a spine CT
  Interventions: Diagnostic Test: 3D spine CT

INTERVENTIONS:
Diagnostic Test: 3D spine CT — CT scan of the spine

SUMMARY:
Volume of the paravertebral spaces of the tharic and lumbar regions will be measured.

DETAILED DESCRIPTION:
Paravertebral block is an effective regional anesthesia method and a golden standart technique for various operations. In addition, paravertebral block is a volume dependent technique. However, there are few cadaveric studies that investigates the volume of the paravertebral space.

This study aims to calculate the volume of the paravertebral spaces of the lumbar and thoracic regions in the patients who had 3D computerized scan in Kocaeli University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had a CT scan of the spine in our hospital

Exclusion Criteria:

* Patients with scoliosis or known vertebral abnormalities

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who had a spine CT scan in our hospital due to vertebral disc degenerative disease
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Lumbar paravertebral space | Baseline
  Volume of the paravertebral space of the lumbar region
Thoracic paravertebral space | Baseline
  Volume of the paravertebral space of the thoracic region

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University Hospital, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No